CLINICAL TRIAL: NCT05711108
Title: Continuous Glucose Monitoring (CGM) to Assess Hypoglycemia in Older Adults With Diabetes in Long Term Care (LTC) Facilities
Brief Title: Continuous Glucose Monitoring (CGM) in Long Term Care (LTC) Facilities
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Collaborators: Theoria Medical (Unknown)
Responsible Party: Sponsor
Other Study IDs: STUDY00000128
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Diabetes; Hypoglycemia; Aging
Keywords: older adults; hypoglycemia; continuous glucose monitoring; long-term care facilities
MeSH Terms: conditions — Diabetes Mellitus; Hypoglycemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Long Term Care Residents Using Glucose Lowering Medication

SUMMARY:
To prospectively determine the burden of hypoglycemia (minutes spent below 70 mg/dl per day, measured by continuous glucose monitor (CGM)) among residents of long term care facilities (LTC) with a diagnosis of type 1 or type 2 diabetes including key clinical subgroups (living in skilled nursing facility (SNF) or nursing home (NH), on different hypoglycemic medications).

This aim will be achieved by recruiting 300 residents with diabetes in 4 LTC facilities. All participants will undergo masked CGM for 10 days.

ELIGIBILITY:
Inclusion Criteria:

* Adults >64 years with diagnosis of type 1 or type 2 diabetes
* Using glucose-lowering medication or insulin

Exclusion Criteria:

* Currently taking or planning to take hydroxyurea
* Patient or Health care proxy refuses to sign consent form

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Long term care residents using glucose lowering medications
Sampling Method: Probability Sample
Enrollment: 86 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Biochemical hypoglycemia | Baseline
  minutes per day sensor glucose <70 mg/dL

SECONDARY OUTCOMES:
A1C | Baseline
Time-in-range | Baseline
  percent/day over 10 days of glucose value between 90-180 mg/dl or 90-250 mg/dl depending current ADA recommendations)
Clinically significant hypoglycemia | Baseline
  minutes per day sensor glucose <54 mg/dl
Severe hypoglycemia | Baseline
  needing 3rd party assistance
Falls, hospitalization | Baseline
Symptoms of hypoglycemia reported to the staff by the resident in between or at the time of fingerstick glucose monitoring (information derived from nursing notes) | Baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided